CLINICAL TRIAL: NCT03977792
Title: A Randomized, Open Label, Non-inferiority Study to Compare the Safety and Efficacy of BOR15001L7 to Docosanol 10% in Patients With Recurrent Herpes Labialis
Brief Title: An Open Label Study to Evaluate the Safety and Efficacy of BOR15001L7 for the Treatment of Cold Sores in Patients With Recurrent Herpes Labialis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratoire Boreaderme Inc. (Industry)
Collaborators: Ecogene 21 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOR-15001L7-P2
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Recurrent Herpes Labialis
Keywords: Herpes Simplex; Skin Diseases, Infectious; Herpesviridae Infections
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex; Skin Diseases, Infectious; Herpesviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental treatment (Experimental): Subjects treated with BOR15001L7.
  All subjects will be randomized 1:1 (BOR15001L7:docosanol 10%) to receive either BOR15001L7 or docosanol 10%.
  Interventions: Drug: BOR15001L7
- Comparator treatment (Active Comparator): Subjects treated with Docosanol 10%.
  All subjects will be randomized 1:1 (BOR15001L7:docosanol 10%) to receive either BOR15001L7 or docosanol 10%.
  Interventions: Drug: Docosanol Cream 10%

INTERVENTIONS:
Drug: BOR15001L7 — BOR15001L7 topically applied to infected area, 5 times a day, until complete healing of the infection.
  Arms: Experimental treatment
Drug: Docosanol Cream 10% — Comparator product topically applied to infected area, 5 times a day, until complete healing of the infection.
  Arms: Comparator treatment

SUMMARY:
BOR15001L7 is a natural product. The primary objective of this study is to demonstrate its non-inferiority to docosanol 10% based on the healing time of cold sores in patients with recurrent herpes labialis.

DETAILED DESCRIPTION:
Secondary objectives are to:

1. Evaluate the efficacy of BOR1500L7 on:

   * The reduction of ulcerative lesions rates following the prodromal stage;
   * The extension of the delay prior to first ulcerative lesions occurence following the prodromal stage;
   * The decrease of cumulative ulcerative lesions dimensions during papule, vesicles, ulcers/soft and hard crust stages;
   * The decrease of symptoms intensity (pain, tingling, itching, burning sensation) during prodromal, erythema, papule, vesicles, ulcers/soft crust, hard crust, re-epithelialize stages;
   * The reduction of symptoms duration (pain, tingling, itching, burning sensation) during the prodromal, erythema, papule, vesicles, ulcers/soft crust, hard crust, re-epithelialize stages in subjects with recurrent herpes labialis;
2. Evaluate the safety and tolerability of BOR15001L7 in subjects with recurrent herpes labialis

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent and willing to comply with study-related procedures;
* Males and females ≥18 years of age at screening;
* Diagnosed with recurrent herpes labialis, defined as showing at least 2 episodes of infections per year;
* Willing to avoid, during the treatment phase, the use of anti-inflammatory, anti-herpetic, antibiotic and antiviral agents as well as steroids or other natural products that would interfere with the immune system response (exception: only the use of valacyclovir will be permitted, if prescribed);
* Willing to avoid, during the treatment phase, the use of cosmetic products (ex. cream, make-up, etc.) at areas close to the infected region.

Exclusion Criteria:

* Patients with skin disease affecting the peribuccal region (eczema, psoriasis, dermatitis, etc.);
* Patients with herpes labialis occurring within 14 days prior to screening;
* Patients known for allergies or intolerance to drug and comparator ingredients, or any cream used to treat skin conditions;
* Treatment with an investigational product or biological agent or device within 30 days or five half˗lives, whichever is longer.
* Any other condition, which, in the opinion of the investigator or the sponsor would make the patient unsuitable for inclusion, or could interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The mean change of healing time | Day 1 to 12

SECONDARY OUTCOMES:
The change in lesion rates following the prodromal stage | Day 1 to 12
The mean change in delays (hours) between the prodromal stage and the first visible occurence of lesions | Day 1 to 12
The percentage change in number of lesions at papule, vesicles and ulcers/soft crust, hard crust stages | Day 1 to 12
The percentage change in dimensions (mm) of lesions at papule, vesicles and ulcers/soft crust, hard crust stages | Day 1 to 12
The percentage of patients that demonstrated a change in intensity of drug-related symptoms (pain, tingling, itching, burning sensation) at papule, vesicles and ulcers/soft crust, hard crust stages | Day 1 to 12
The mean change in duration (hours) of drug-related symptoms (pain, tingling, itching, burning sensation) at papule, vesicles and ulcers/soft crust, hard crust stages | Day 1 to 12
Safety and tolerability measured by the Incidence of Treatment-Emergent Adverse Events [Side-effects] | Day 1 to 12

REFERENCES:
- [Background] Lavoie S, Cote I, Pichette A, Gauthier C, Ouellet M, Nagau-Lavoie F, Mshvildadze V, Legault J. Chemical composition and anti-herpes simplex virus type 1 (HSV-1) activity of extracts from Cornus canadensis. BMC Complement Altern Med. 2017 Feb 22;17(1):123. doi: 10.1186/s12906-017-1618-2. PMID 28228101